CLINICAL TRIAL: NCT01032343
Title: The Effect of Omega-3 Polyunsaturated Fatty Acids on UV-induced Immunosuppression
Brief Title: An Immunonutritional Approach to the Prevention of Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Lesley Rhodes, Professor of Experimental Dermatology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AICR 08-0131; UKCRN 6873 (Registry Identifier: UK Clinical Research Network)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Skin Cancer
Keywords: Immunosuppression; Ultraviolet radiation; Nickel; Contact hypersensitivity
MeSH Terms: conditions — Skin Neoplasms; Dermatitis, Contact | interventions — Docosahexaenoic Acids; Gelatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 PUFA capsule (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 PUFA
- Gelatine capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Gelatine

INTERVENTIONS:
Dietary Supplement: Omega-3 PUFA — One capsule (4g omega-3 PUFA) daily for 3 months
  Arms: Omega-3 PUFA capsule
Dietary Supplement: Gelatine — One capsule daily for 3 months
  Arms: Gelatine capsule

SUMMARY:
Skin cancer incidence continues to rise and ultraviolet radiation (UVR) in sunlight is the principal cause. Solar UVR can promote cancer development through its ability to suppress the immune system. The purpose of this study is to determine whether dietary supplementation with omega-3 polyunsaturated fatty acids can protect human skin from UVR-induced immunosuppression.

DETAILED DESCRIPTION:
Skin cancer is one of the most common human cancers with a rising incidence and considerable negative impact on human health. Exposure to ultraviolet radiation (UVR) in sunlight is the major aetiological factor in skin cancer initiation and progression. Human case-control studies have reported an inverse relationship between dietary fish or omega-3 polyunsaturated fatty acid (PUFA) intake and occurrence of non-melanoma skin cancer. Omega-3 PUFA have the potential to reduce the risk of photocarcinogenesis primarily by their ability to reduce production of prostaglandin E2 and consequently photoimmunosuppression. To date, no studies have assessed the impact of omega-3 PUFA on skin photoimmunosuppression in humans.

OBJECTIVE: To examine the potential of dietary omega-3 PUFA to protect against UVR-induced cutaneous immunosuppression in humans.

STUDY DESIGN: A double-blind randomised controlled nutritional study in 64 healthy human volunteers with nickel sensitivity. Volunteers will receive 3 months dietary supplementation with either omega-3 PUFA (n=32) or gelatine (n=32) both provided in identical gelatine capsules.

The aim is to quantify the influence of omega-3 PUFA on:

1. UVR-induced suppression of clinical contact hypersensitivity (CHS) responses
2. UVR-induced modulation of epidermal Langerhans cell trafficking
3. UVR-induced modulation of levels of immunoregulatory mediators

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females
* Sun-reactive skin type I / II
* Reporting allergy to jewellery with nickel content

Exclusion Criteria:

* History of atopy
* History of skin cancer
* History of a photosensitivity disorder
* Sunbathing (including sunbeds) in the last 3 months
* Pregnancy
* History of cardiac disease
* Taking photoactive medicine
* Not able to eat fish or gelatine
* Taking fish oil supplements prior to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Degree of suppression of nickel-induced contact hypersensitivity | 3 months
  Measurement of the erythema of nickel-induced eczema using a reflectance instrument

SECONDARY OUTCOMES:
Intergroup comparison of cytokine and eicosanoid levels and Langerhans cell numbers | 3 months
Correlation of susceptibility to photoimmunosuppression in all subjects with their erythrocyte omega-3:omega-6 PUFA ratio | 3 months
Correlation of susceptibility to photoimmunosuppression with cytokine and eicosanoid levels and Langerhans cell numbers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lesley E Rhodes, MBBS, MD, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Result] Pilkington SM, Massey KA, Bennett SP, Al-Aasswad NM, Roshdy K, Gibbs NK, Friedmann PS, Nicolaou A, Rhodes LE. Randomized controlled trial of oral omega-3 PUFA in solar-simulated radiation-induced suppression of human cutaneous immune responses. Am J Clin Nutr. 2013 Mar;97(3):646-52. doi: 10.3945/ajcn.112.049494. Epub 2013 Jan 30. PMID 23364005
- [Derived] Pilkington SM, Rhodes LE, Al-Aasswad NM, Massey KA, Nicolaou A. Impact of EPA ingestion on COX- and LOX-mediated eicosanoid synthesis in skin with and without a pro-inflammatory UVR challenge--report of a randomised controlled study in humans. Mol Nutr Food Res. 2014 Mar;58(3):580-90. doi: 10.1002/mnfr.201300405. Epub 2013 Dec 5. PMID 24311515
- See also: Study recruitment information — http://www.staffnet.manchester.ac.uk/volunteering/display/index.htm?id=149716